CLINICAL TRIAL: NCT07334847
Title: Efficacy of Anterior Foot Wedge Modulation With Neuromuscular Training on Balance During Walking in Parkinsonian Patients
Brief Title: Anterior Foot Wedge With Neuromuscular Training for Balance in Parkinson's Disease
Acronym: AFW-NT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, reda abd elrazik, Associate Professor of Physical Therapy, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PT. BU. EC. 29
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease; Postural Instability; Gait Disorder
Keywords: Anterior foot wedge; Neuromuscular training; Balance; Gait; Biodex; Electromyography; Postural stability
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: "Two-group randomized controlled trial comparing conventional physical therapy (control) versus conventional therapy plus anterior foot wedge and neuromuscular training (experimental)."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Training + Anterior Foot Wedge + Conventional PT (Experimental): Participants will receive a 60-minute session, 3 times per week for 8 weeks, consisting of: (1) conventional physical therapy including proprioceptive neuromuscular facilitation (PNF) for head, neck, and trunk; stretching of lower limb flexors; strengthening of lower limb extensors and trunk muscles; and balance/weight-shifting exercises; (2) a customized anterior foot wedge worn during all training sessions to modulate center of pressure; and (3) neuromuscular training using the Biodex Multi-Joint System to enhance postural control and gait stability.
  Interventions: Device: Anterior foot wedge; Behavioral: Neuromuscular training
- Conventional Physical Therapy Only (Active Comparator): articipants will receive a 60-minute session, 3 times per week for 8 weeks, consisting of conventional physical therapy including: proprioceptive neuromuscular facilitation (PNF) for head, neck, and trunk; stretching of lower limb flexor muscles; strengthening of lower limb extensor and trunk muscles; balance exercises; and weight-shifting and gait training.
  Interventions: Behavioral: Neuromuscular training

INTERVENTIONS:
Device: Anterior foot wedge — A custom-made orthotic insert placed under the forefoot to shift the center of pressure anteriorly, thereby enhancing postural stability and balance during walking and standing tasks in Parkinsonian patients.
  Arms: Neuromuscular Training + Anterior Foot Wedge + Conventional PT
Behavioral: Neuromuscular training — A structured training program using the Biodex Multi-Joint System to improve dynamic balance, motor control, and gait stability through reactive and perturbation-based exercises, performed 3 times per week for 8 weeks.

SUMMARY:
This study will test whether combining an anterior foot wedge with neuromuscular training can improve balance, gait, and muscle activity in people with Parkinson's disease. Thirty patients (ages 45-75) with moderate Parkinson's (Hoehn & Yahr Stage III) will be randomly assigned to one of two groups:

Group 1 (Control): Receives a standard physical therapy program including stretching, strengthening, PNF, weight-shifting, and gait training.

Group 2 (Experimental): Receives the same physical therapy plus neuromuscular training using the Biodex Multi-Joint System and a custom anterior foot wedge.

All participants will train for 60 minutes, three times per week, for 8 weeks. Before and after the program, researchers will measure: balance (using the Biodex Balance System), gait (via Unified Parkinson's Disease Rating Scale and motion analysis), and muscle activity in the trunk (using electromyography). The goal is to find a more effective rehabilitation approach to reduce fall risk and improve walking in Parkinson's patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease, confirmed by neurologist. Disease severity classified as Stage III on the Hoehn & Yahr scale. Age between 45 and 75 years. Medically stable (normal vital signs). Conscious, cooperative, and able to follow instructions. No severe cognitive or psychological impairment. Able to provide informed consent.

Exclusion Criteria:

* Severe disability or advanced Parkinsonism (Stage IV or V). Presence of other neurological or orthopedic conditions affecting gait or balance (e.g., stroke, spinal cord injury, severe arthritis).

History of diabetes in second-degree relatives (as specified in your protocol). Unstable medical conditions (e.g., uncontrolled hypertension, cardiac disease). Inability to stand or walk with minimal assistance. Non-cooperative or unable to tolerate assessment procedures (EMG, Biodex, motion analysis).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Change in Limit of Stability (LOS) | Baseline and after 8 weeks of intervention (24 sessions)
  Measured using the Biodex Balance System SD (Model BLS003, USA). The Limit of Stability test assesses the patient's ability to voluntarily shift their center of gravity to the maximum distance in eight directions without losing balance. Results are reported as a composite stability index score (lower = better stability).

SECONDARY OUTCOMES:
Change in Gait Disability (UPDRS Score) | Baseline and after 8 weeks
  Assessed using Part III (Motor Examination) of the Unified Parkinson's Disease Rating Scale (UPDRS), specifically items related to gait, posture, and postural stability. Total score ranges from 0 (no disability) to higher values (greater impairment).
Change in Step Length | Baseline and after 8 weeks
  Measured using a 3D motion analysis system (Hocoma, Model 000341, USA). Average step length (distance between successive heel strikes) in centimeters during comfortable walking speed.
Change in Walking Velocity | Baseline and after 8 weeks
  Measured via motion analysis system during a 10-meter walk test. Reported in meters per second.
Change in Cadence | Baseline and after 8 weeks
  Number of steps per minute during walking, recorded by motion analysis system.
Change in Electromyographic (EMG) Amplitude of Trunk Muscles | Baseline and after 8 weeks
  Surface EMG (Neuropac S1, Model DI 90B, Japan) used to record amplitude of motor unit action potentials (in microvolts, µV) from rectus abdominis and erector spinae muscles during standing and walking tasks.

IPD SHARING:
Plan to Share IPD: Undecided